CLINICAL TRIAL: NCT05403268
Title: The Impact of Early Delirium Detection With DeltaScan on Management of Underlying Delirium Causes in Critically Ill Patients. A Randomized Controlled Trial.
Brief Title: The EARLY DELTA Trial
Acronym: EARLY DELTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Ottens (Other)
Collaborators: Prolira (Industry); Dutch Society of Intensive Care (Unknown)
Responsible Party: Sponsor-Investigator, Thomas Ottens, Consultant Anesthesiologist-Intensivist, HagaZiekenhuis
Organization: HagaZiekenhuis (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: T21-064; NL78854.041.21 (Registry Identifier: CCMO Toetsingonline)
Record Dates: First submitted 2022-05-13; First posted 2022-06-03 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Delirium; Critical Illness; Acute Encephalopathy
Keywords: acute encephalopathy; delirium; critical illness; intensive care unit; automated EEG; electroencephalography
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 parallel arms: control group (usual care) and intervention group.
Masking Description: Usual care group undergoes DeltaScan measurements with blinded device to prevent the measurement result from influencing clinical decisions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Sham Comparator): Usual care group. Participants undergo twice daily DeltaScan measurements in addition to usual care. An adapted device is used, that masks the measurement result (it generates a QR-code, that is scanned into the patient data management system). The results will be unblinded one enrollment is complete.
  Interventions: Device: DeltaScan
- Usual Care + DeltaScan (Experimental): Intervention group. Participants undergo twice daily DeltaScan measurements in addition to usual care. The measurement result is used together with routine delirium screening observations to guide management, according to the local delirium protocol.
  Interventions: Device: DeltaScan

INTERVENTIONS:
Device: DeltaScan — Twice daily DeltaScan observations
  Other Names: automated 1-channel EEG

SUMMARY:
Rationale: Delirium is a type of acute encephalopathy that is triggered by an underlying somatic disorder. Patients experience disturbances in attention, alertness and other cognitive functions. In patients with delirium, a characteristic electroencephalography (EEG) pattern is seen, known as polymorphic delta activity. The MDR certified medical device "Deltascan" can detect this EEG pattern. Traditional clinical delirium screening instruments are known to have limited sensitivity, in particular for detecting hypoactive delirium. We hypothesize that adding EEG based encephalopathy detection to clinical observation scales increases the sensitivity and results in earlier detection of delirium and subsyndromal delirium, resulting in improved clinical outcomes of critically ill patients, such as delirium duration, ICU length of stay or survival.

Objective: This randomized controlled trial aims to study the effect of implementation of EEG based encephalopathy detection (DeltaScan, Prolira, Utrecht, The Netherlands, hereafter: DeltaScan) on relevant clinical endpoints (ICU length of stay, sedative requirements and delirium related complications, among others) in a mixed medical and surgical intensive care unit population.

Study design: a randomized controlled trial Study population: adult patients (>18 years) admitted to the ICU for unplanned care with a minimal anticipated ICU length of stay of 48h.

Intervention: either usual care, where the patients' medical team obtains regular delirium screening, versus usual care plus twice daily DeltaScan measurements. During the daily medical rounds, the DeltaScan results will be presented to the patients' medical team together with decision support, consisting of DeltaScan trend interpretation and protocol-based suggestions for evaluation of underlying delirium cause.

Main study parameters/endpoints: primary endpoint will be ICU length of stay. Secondary endpoints are encephalopathy/delirium occurrence, ICU encephalopathy/delirium free days, ventilator free days, organ support free days, sedative, opioid and antipsychotic drug requirement, delirium related complication occurrence, frequency and duration of physical restraints application, ICU mortality, ICU readmission, hospital length of stay, hospital mortality and 90-day mortality.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In this study, it is not expected that randomization to the intervention group adds risk for patients. This is a study of a diagnostic intervention with additional encephalopathy/delirium observations consisting of a short (90 seconds) EEG measurement, which does not harm the patient. Clinicians will receive protocol-based decision support alongside the diagnostic observation. No additional medical treatments will be conducted as part of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or above) admitted to ICU for any indication
* ICU length of stay anticipated to be 48h or longer from time of screening for inclusion
* Written informed consent by patient or representative

Exclusion Criteria:

* More than 48 hours have elapsed since the patient was first eligible to undergo a DeltaScan measurement after ICU admission. A patient is eligible for DeltaScan measurements if they are a. able to cooperate with simple instructions AND b. are alert or mildly sedated no deeper than a Richmond Agitation and Sedation Score of -2.
* Admission for out-of-hospital cardiac arrest, status epilepticus, hemorrhagic or ischemic stroke, increased intracranial pressure, head trauma
* Recent intracranial neurosurgery (<30 days prior to inclusion)
* Known space-occupying lesions in the brain or skull
* Metal implants in brain or skull
* Diagnosis of dementia or Parkinson's disease
* Inpatient from nursing home
* Lithium use (<30 days prior to inclusion)
* Imminent death or palliative care phase
* Patients ánd their legal representatives both do not understand Dutch or English
* Patients who participated in the EARLY DELTRA trial <90 days ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
ICU length of stay | Assessed at the 90 day post discharge follow-up
  Length of stay in the intensive care unit, measured in hours

SECONDARY OUTCOMES:
Encephalopathy/delirium occurrence (DeltaScan) | Assessed daily, until participant is discharged from ICU, or until the maximum observation time (30 days)
  Defined as: any DeltaScan score ≥ 3 OR initiation of antipsychotic treatment
Delirium occurrence (ICDSC) | Assessed daily, until participant is discharged from ICU, or until the maximum observation time (30 days)
  Defined as: any ICDSC score ≥ 4 OR initiation of antipsychotic treatment
ICU encephalopathy/delirium and coma free days (reported as: composite, delirium free days, coma free days) | Assessed at the 14th day after ICU admission. If the patient dies during the first 14 days of the study observation period, this outcome is assessed at the date of death
  Defined as: the number of days in the first 14 days after the patient was randomized during which the patient was alive without delirium or coma. We will calculate this value separately based on DeltaScan alone, DeltaScan+ICDSC and ICDSC alone)
ICU ventilator free days | Assessed at the 14th day after ICU admission. If the patient dies during the first 14 days of the study observation period, this outcome is assessed at the date of death
  Defined as: the number of days in the first 14 days after the patient was randomized during which the patient was alive without mechanical ventilation, regardless of ventilation mode or route. High-flow nasal oxygen (HFNO) will not be regarded as ventilation. If patients are ventilated with a device provided by another institute (i.e. Centrum voor Thuisbeademing), only days spent on the ICU ventilator will be counted. Any day with <12h of mechanical ventilation will be counted as 0,5 day. More than 12h of mechanical ventilation will be counted as 1 day
ICU organ support free days | Assessed at the 14th day after ICU admission. If the patient dies during the first 14 days of the study observation period, this outcome is assessed at the date of death
  Defined as: the number of days in the first 14 days after the patient was randomized during which the patient was alive without mechanical ventilation (any modality), HFNO, renal replacement therapy (any modality), mechanical circulatory support (ECLS, IABP, Impella), intravenous inotropes (dobutamine, milrinone, enoximone, levosimendan) or vasopressors (noradrenalin > 0.25 mcg/kg/min or any dose of terlipressin / arginine vasopressin)
ICU mortality rate | This is assessed at the date of death. In ICU survivors, it is assessed at the 90 day post-discharge follow-up
  Defined as death occurring before ICU discharge. Outcome reported as proportion of participants who died before ICU discharge.
ICU readmission rate | This outcome is only scored when an unplanned re-admission occurs within the first 90 days after ICU discharge.
  Unplanned re-admission to the ICU before hospital discharge. Outcome reported as proportion of participants who were re-admitted to ICU before hospital discharge.
Hospital length-of-stay | Assessed at the 90 day post-discharge follow-up
  Outcome reported in days
Hospital mortality rate | This is assessed at the date of death. In survivors, it is assessed at the 90 day post-discharge follow-up
  Defined as death occurring before hospital discharge. Outcome reported as proportion of participants who died before hospital discharge.
90 day mortality rate | Assessed at the 90 day post-discharge follow-up
  Defined as death occurring within 90 days after study enrollment. Outcome reported as proportion of participants who died before 90d follow-up
ICU Sedative Drug requirement | Assessed daily, until participant is discharged from ICU, or until the maximum observation time (30 days)
  The cumulative doses of the following sedative drugs, administered after randomisation: propofol, clonidine, dexmedetomidine, esketamine, zopiclone, benzodiazepines
ICU opioid requirement | Assessed daily, until participant is discharged from ICU, or until the maximum observation time (30 days)
  The cumulative doses of opioids, administered after randomisation
ICU antipsychotic drug requirement | Assessed at ICU Assessed daily, until participant is discharged from ICU, or until the maximum observation time (30 days)
  cumulative dose of the following antipsychotic drugs, administered after randomisation: haloperidol, quetiapine, other antipsychotic drugs
ICU accidental device removal incidence and falls | Assessed daily, until participant is discharged from ICU, or until the maximum observation time (30 days)
  Defined as the number of incidents where a patient accidentally removes an indwelling catheter, tube, infusion line or drain (e.g. intravenous lines, wound drains, airway device, feeding tubes etc) or falls out of bed
ICU incidence and duration of the use of physical restraints | Assessed daily, until participant is discharged from ICU, or until the maximum observation time (30 days)
  Defined as the frequency of application of physical restraints and the cumulative duration of restraint application during ICU admission
Self-assessed quality of life | Assessed one year after ICU discharge
  Self-assessed quality of life measured with the Euroqol Quality of Life questionnaire, version EQ6D
Self assessed cognitive function | Assessed one year after ICU discharge
  Self-assessed cognitive function measured with the cognitive failure questionnaire (CFQ, Merckelbach, Muris & Nijman 1996)
Self assessed mood and depression symptoms | Assessed one year after ICU discharge
  Self assessed mood and depression symptoms measured with the Patient Health Questionnaire (PHQ-9)
Self assessed mobility and physical functioning | Assessed one year after ICU discharge
  Self assessed mobility and physical functioning measured with the Barthel Index

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Ottens, MD, MSc, PhD, Principal Investigator — HagaZiekenhuis
Locations (2):
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede, Overijssel
  - HagaZiekenhuis, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: No